CLINICAL TRIAL: NCT04707742
Title: Clinical Evaluation of Antiseptic Mouth Rinses to Reduce Salivary Viral Load of SARS-CoV-2 in COVID-19 Patients
Brief Title: Antiseptic Mouth Rinses to Reduce Salivary Viral Load in COVID-19 Patients
Acronym: BUCOSARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Collaborators: Hospital Universitario Fundación Jiménez Díaz (Other); Hospital Universitario General de Villalba (Unknown); Hospital Universitario Infanta Elena (Unknown); Hospital Universitario Virgen de la Arrixaca (Other); Hospital Clínico Universitario de Valencia (Other); Dentaid SL (Industry)
Responsible Party: Principal Investigator, Alejandro Mira Obrador, BSc in Biological Sciences (Alicante University), MSc PhD (Oxford University), Senior Researcher (FISABIO Foundation), Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Interventional
Record Dates: First submitted 2021-01-07; First posted 2021-01-13 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-09

CONDITIONS: Covid19
Keywords: COVID-19; MOUTHWASHES; SALIVA; VIRAL LOAD; ORAL; CLINICAL TRIAL
MeSH Terms: conditions — COVID-19 | interventions — Povidone-Iodine; Hydrogen Peroxide; Cetylpyridinium

STUDY DESIGN:
Intervention Model Description: A multicentre, randomized, blind, five-parallel-group, placebo-controlled trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The hospital staff consecutively assigned each participant a code following the order from a previously randomly generated table.
  The code were unknown to the personnel who processed the samples and to those that analyzed the data.
  Participants were blinded by using identical tubes with the same volume for both mouthwashes and placebo.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Povidone-iodine 2% (Betadine© bucal 100 mg/ml) (Experimental): Povidone-iodine 2% (Betadine© bucal 100 mg/ml) (Mylan Pharmaceuticals, S.L., Spain).
  The concentration was adjusted to those previously indicated by diluting commercial formulas with distilled water minutes before rinsing (3 mL of povidone-iodine 10% for oral use - Betadine© with 12 mL of distilled water).
  Interventions: Drug: Betadine© bucal 100 mg/ml
- Hydrogen peroxide 1% (Oximen® 3%) (Experimental): Hydrogen peroxide 1% (Oximen® 3%) (Reig Jofré, S.A., Spain). The concentration was adjusted to those previously indicated by diluting commercial formulas with distilled water minutes before rinsing (5 mL of hydrogen peroxide 3% - Oximen© with 10 mL of distilled water).
  Interventions: Drug: Oximen® 3%
- Clorhexidine 0,12% (Clorhexidine Dental PHB©) (Experimental): Clorhexidine 0,12% (Clorhexidine Dental PHB©) contains clorhexidine (C22H30N10Cl2).
  Rinses were ready to use in their commercial formulas.
  Interventions: Drug: Clorhexidine Dental PHB©
- Cetylpyridinium chloride 0,07% (Vitis Xtra Forte©) (Experimental): Cetylpyridinium chloride 0,07% (Vitis Xtra Forte©) contains cetylpyridinium chloride (C21H38ClN).
  Rinses were ready to use in their commercial formulas.
  Interventions: Drug: Vitis Xtra Forte©
- Control (Distilled Water) (Placebo Comparator): Distilled water.
  Interventions: Drug: Distilled Water

INTERVENTIONS:
Drug: Betadine© bucal 100 mg/ml — 15 ml 2% povidone-iodine, one minute rinse.
  Other Names: Povidone-iodine
  Arms: Povidone-iodine 2% (Betadine© bucal 100 mg/ml)
Drug: Oximen® 3% — 15 ml 1% hydrogen peroxide, one minute rinse.
  Other Names: H2O2; Hydrogen peroxide
  Arms: Hydrogen peroxide 1% (Oximen® 3%)
Drug: Clorhexidine Dental PHB© — 15 ml 0,12% clorhexidine, one minute rinse.
  Other Names: C22H30N10Cl2
  Arms: Clorhexidine 0,12% (Clorhexidine Dental PHB©)
Drug: Vitis Xtra Forte© — 15 ml 0,07% cetylpyridinium chloride, one minute rinse.
  Other Names: C21H38ClN; Cetylpyridinium chloride
  Arms: Cetylpyridinium chloride 0,07% (Vitis Xtra Forte©)
Drug: Distilled Water — 15 ml distilled water, one minute rinse.
  Other Names: H2O
  Arms: Control (Distilled Water)

SUMMARY:
As no curative treatment for SARS-CoV-2 is currently available, most public health measures to contain the pandemic are based on preventing the spread of the pathogen. The virus is transmitted by the respiratory route and by direct contact with contaminated surfaces and subsequent contact with nasal, oral or ocular mucosa. Although patients with symptomatic coronavirus disease 2019 (COVID-19) have been the main source of transmission, observations suggest that asymptomatic and incubating patients also have the ability to transmit SARS-CoV-2. Angiotensin II converting enzyme (ACE2) is the main cellular receptor for SARS-CoV-2, which interacts with the spike protein to facilitate its entry. ACE2 receptors are highly expressed in the oral cavity and present at high levels in oral epithelial cells. The mean expression of ACE2 was higher in the tongue compared to that in other oral tissues and it has been found to be higher in the minor salivary glands than in the lungs. These findings strongly suggest that the oral cavity and specifically the saliva may be a high-risk route for SARS-CoV-2 infection. Thus, strategies reducing salivary viral load could contribute to reduce the risk of transmission. Furthermore, studies using macaques as animal models have shown that SARS-CoV persists for two days in oral mucous membranes before its diffusion to the lower respiratory tract. This offers an interesting preventive and therapeutic window of opportunity for the control of this disease. For this reason, the use of mouthwashes with antiseptics that have virucidal activity can be a simple preventive strategy that could easily be applied both by infected patients before being examined by sanitary personnel and in the general population. This study is a multi-centered, blinded, parallel-group, placebo-controlled randomised clinical trial that tests the effect of four different mouthwashes (CPC, chlorhexidine, povidone-iodine and H2O2) in the salivary viral load of SARS-CoV-2 measured by qPCR at three different timepoints. A fifth group of patients using a distilled water mouth rinse is used as a control. Viral particles per ml of saliva are quantified at baseline and 30, 60 and 120 minutes after a 1-minute mouth rinse with the antiseptic or water. Our study aims to test whether any of these standard oral antiseptics appear to diminish viral load in saliva and could therefore be used as a strategy to reduce transmission risk in clinical and social settings.

DETAILED DESCRIPTION:
Strategies reducing salivary viral load could contribute to reduce the risk of transmission of SARS-CoV-2. Thus, the use of mouthwashes with antiseptics that have virucidal activity can be a simple and low-cost preventive strategy that could easily be applied in the general population. To evaluate the effect of several antiseptics to neutralize or reduce the SARS-CoV-2 viral load in vivo in saliva samples, a multicentre, randomized, blind, five-parallel-group, placebo-controlled trial has been designed.

The study will be performed in Madrid, Valencia and Murcia regions in Spain, in five different hospitals: Fundación Jiménez Díaz University Hospital (Madrid, Spain), Villalba University General Hospital (Madrid, Spain), Infanta Elena University Hospital (Madrid, Spain), Virgen de la Arixaca University Hospital (Murcia, Spain) and Clínico de Valencia University Hospital (Valencia, Spain).

Every patient included is previously diagnosed and hospitalized because of SARS-COV-2 infection, being admitted mainly for respiratory pathology. All of them will be adults (age >18 years) and provide their voluntary written or oral consent to participation according to the hospital's ethics committee recommendations.

After approval of consent, the hospital staff responsible for the interventions will consecutively assign each participant a code following the order from a previously randomly generated table. The code will consist of a patient number and a letter corresponding to one of the five study groups (A, B, C, D and E), that will be known to the clinical personnel but unknown to the laboratory personnel who will process samples and extract RNA, as well as to those that will analyse the data. In this way, participants will be randomly assigned to one of the five treatment groups and the blind will be achieved by using identical tubes with the same volume for both mouthwashes and placebo.

Every included patient is asked not to eat, drink anything but water, chew gum, smoke, brush their teeth, or use any mouthwash for one hour prior to sample collection. In addition, they are not allowed to drink for half an hour after the mouthwash and eat for the entire test.

Five mouthwashes are randomized: 2% povidone-iodine (group A), 1% hydrogen peroxide (group B), 0.12% chlorhexidine (group C), 0.07% cetylpyridinium chloride (group D) and distilled water (group E), as the control group. Group C (Clorhexidina dental PHB©) and D (Vitis Xtra Forte©) rinses are ready to use in their commercial formulas. In the case of the mouthwashes A and B, the concentrations have to be adjusted to those previously indicated by diluting commercial formulas with distilled water minutes before rinsing (3 mL of povidone-iodine 10% for oral use with 12 mL of distilled water, in group A; and 5 mL of hydrogen peroxide 3%- Oximen© with 10 mL of distilled water, in group B). All mouthwashes and their respective dilutions are commercial products classified as safe.

A total of 4 non stimulated saliva samples will be collected for each patient: one basal and three after the mouthwash, at 30 minutes, at 60 minutes and at 120 minutes, respectively. The patients will be asked to provide each unstimulated saliva sample into a sterile 10 cm diameter plastic container (at least 0.5 mL of sample) by drooling, avoiding spilling secretions of bronchial origin. Immediately after each sampling, 0.5 mL of saliva will be transferred to a sterile Eppendorf tube with 1.5 mL of virus inactivating buffer labeled with the patient code and sample time and kept at 4 °C. The four Eppendorf tubes per patient will be introduced in an airtight bag, containing protecting absorbent material in case of undesired opening or breaking. The secondary containers will be introduced in a rigid box according to UN3733 standards and sent to laboratory by courier service for analysis.

An aliquot of 1 ml of each saliva sample diluted in the virus inactivating buffer in proportion 1:3, will be used for RNA extraction using a standard TRIzol-based method. Briefly, 3 ml of TRIzol and 600 ul of chloroform will be added, vortexed vigorously for 15 seconds and incubated on ice for 10 minutes. Then, samples will be centrifuged at 12,000 g for 15 min at 4 °C and the aqueous phase transferred to two clean microtubes with 750 ul of isopropanol. Tubes will be mixed by inversion and incubated during 15 minutes before centrifugation at 12,000 g for 10 minutes at 4 °C. Supernatant will be discarded by decantation and pellets washed with 1 ml 80% cold ethanol, vortexed to mix thoroughly and centrifugated at 7,500 g for 5 minutes at 4 °C. Supernatants will be carefully aspirated and discarded, and pellets dried at room temperature for 10 minutes before being resuspended in 15 ul of RNAse -free water and pooled in a single tube.

One step rRT-PCR will be performed using SuperScript™ III One-Step RT-PCR System with Platinum™ Taq DNA Polymerase (Invitrogen-12574026) according to manufacturer's instructions. For the amplification of the SARSCoV-2 E (betacoronavirus screening assay) gene, PCR will be performed following the Charité-Berlin protocol in a LightCycler 480 2.0 (Roche) platform. In the same run, samples will be amplified with housekeeping human gene RNP (Ribonuclease P) primers to assess specimen quality. All samples will be run in two replicates, together with a previously known positive and negative controls. Virus copies will be quantified using a 10-fold dilution standard curve of RNA transcripts previously generated (EDX SARS-CoV-2 Standard, EXACT DIAGNOSTICS EDX). Virus copies were normalized by ml of saliva.

Regarding the analyses to be performed, the main objective of the study is to determine the effect of the different mouthwashes on the SARS-Cov2 viral load in saliva tested in vivo. Thus, the primary outcome will be the change in salivary viral load between baseline and the three post-mouthwash timepoints in each treatment. In addition, the correlations between the basal viral load prior to rinsing with the different clinical data collected, such as age, sex, days since the appearance of symptoms and days since the patients' virus positivity determined by PCR of nasopharyngeal samples will also be studied. Finally, the possible associations between categorical clinical variables and the frequency of patients who improve in viral load at different times for the different treatments will be evaluated.

Considering that each volunteer act as their own control, when comparing the viral load values in saliva at every time with respect to the levels prior to rinsing with the mouthwash, a sample size of 15 patients per branch was considered sufficient to identify significant viral load differences of more than 20% between timepoints, assuming a 10% loss of patients due to abandonment or low viral load and adopting an alpha of 0.05 and a power of 0.8. As 5 branches were programmed in the trial (povidone-iodine, hydrogen peroxide, chlorhexidine, cetylpyridinium chloride and the control), 75 patients were the minimum number of total individuals to be recruited, who will be distributed among the different hospitals.

A Wilcoxon signed-rank test will be used to test average differences, both for the paired case, (when comparing observations in different timepoints for the same individuals), and for the un-paired case (when comparing different treatments based on relative changes of viral load). In addition, some tests for association between paired samples using Spearman's correlation coefficients will be performed to assess the relationship between viral load and other clinical continuous variables. Finally, in order to evaluate associations between clinical categorical variables and the frequency of responders/non-responders to the treatments, the investigators will carry out chi-squared contingency table tests. The investigators define as responder an individual exhibiting an improvement equal to or greater than 90% of basal viral load. All computations and tests will be performed using R environment for statistical computing version 3.6.3 and its 'stats' package [R Core Team 2020].

In addition, to determine the effect of the mouthwashes on the viability of the viruses in saliva, an addendum was submitted to the hospital's ethics committee and after its approval, 62 more patients were recruited for the study. In this case the protocol included a number of modifications, namely: (i) the use of basal, 30 minutes and 60 minutes samples only (2 hour samples excluded); (ii) not using virus inactivating buffer to ensure viral viability; (iii) an in vitro infection assay to determine the infectious capacity of the salivary viruses (infective viral load), which has been included as an additional outcome. The details are described below.

The study will be performed in Madrid, Valencia and Murcia regions in Spain, in four different hospitals: Fundación Jiménez Díaz University Hospital (Madrid, Spain), Villalba University General Hospital (Madrid, Spain), Infanta Elena University Hospital (Madrid, Spain) and Virgen de la Arixaca University Hospital (Murcia, Spain).

A total of 3 non stimulated saliva samples will be collected for each patient: one basal and two after the mouthwash, at 30 minutes and at 60 minutes, respectively. The patients will be asked to provide each unstimulated saliva sample into a sterile 10 cm diameter plastic container (at least 2 mL of sample) by drooling, avoiding spilling secretions of bronchial origin. The three samples will be immediately stored at -80ºC in airtight bags until they are sent to the laboratory. For sample analysis, all secondary containers of airtight bags with the three saliva samples of each patient will be introduced in a rigid box with dry ice according to UN3733 standards and sent to the laboratory (FISABIO) by courier service.

When receiving the samples at the FISABIO Foundation, they will be processed in the facilities of the level 3 security laboratory as follows. After thawing the samples at room temperature, a 200 uL aliquot will be taken for RNA extraction, and the rest will be aliquoted and immediately stored at -80C for assay in cell lines.

RNA extraction will be carried out with the fully automated platform eMAG (bioMérieux, France) following the manufacturer's instructions for saliva samples. One step rRT-PCR and the amplification of the SARSCoV-2 will be performed as described above.

For the cell culture, Vero-E6 cells (ATCC) are cultured in DMEM supplemented with 10% heat-inactivated fetal bovine serum (FBS), 1% Penicillin/Streptomycin (P/S), 1% non-essential amino acids, 1% L-glutamine and 25mM HEPES. All cells are incubated at 37°C and 5% CO2.

Saliva samples will be diluted 1:1 in 1X Dulbecco's PBS. 300 ul of diluted saliva samples will be incubated for one hour at 37°C and 5% CO2 with 1.5x105 Vero-E6 cells in a 24-well plate. Unbound virus will be extracted and the media replaced by 500 ul of infection media (DMEM with 2% FBS, 1% Penicillin/Streptomycin (P/S), 1% non-essential amino acids, 1% L-glutamine, 25mM HEPES and Tripsine TPCK 6ug/ml). Infected Vero-E6 cells will be incubated at 37°C and 5% CO2. After 5 days of infection, supernatant will be collected for RNA extraction following the eMAG platform instructions and one step rRT-PCR performed for the amplification of the SARSCoV-2. The viral load obtained after this 5-day infection period will be considered the infective viral load.

ELIGIBILITY:
Inclusion Criteria:

* Lower than 7 days from the positive SARS-COV-2 PCR test of a nasopharyngeal sample
* Have the ability to donate saliva samples and perform mouthwash

Exclusion Criteria:

* Patient participation in a COVID-19 research study using experimental drugs,
* Use of an antiseptic mouthwash for 48 h before the start of the study
* Any known hypersensitivity or allergy to components of the mouthwashes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-09-18 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Effect of 5 different mouthwashes on the SARS-Cov2 viral load. | Minute 0 (before mouthwash) - Minute 30 (after mouthwash) - Minute 60 (after mouthwash) - Minute 120 (after mouthwash)
  Determine the changes on the SARS-Cov2 viral load in saliva tested in vivo, between baseline values and those obtained at 30 minutes, at 60 minutes and at 120 minutes, after the use of 5 different mouthwashes randomized on 98 COVID-19 patients.
Effect of 5 different mouthwashes on the infective SARS-Cov2 viral load in saliva. | Minute 0 (before mouthwash) - Minute 30 (after mouthwash) - Minute 60 (after mouthwash)
  Determine the changes on the SARS-Cov2 infective viral load in saliva tested in vivo, between baseline values and those obtained at 30 minutes and at 60 minutes after the use of 5 different mouthwashes randomized on 62 COVID-19 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Mira, PhD, Principal Investigator — Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Locations (1):
- Alejandro Mira, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanchez Barrueco A, Mateos-Moreno MV, Martinez-Beneyto Y, Garcia-Vazquez E, Campos Gonzalez A, Zapardiel Ferrero J, Bogoya Castano A, Alcala Rueda I, Villacampa Auba JM, Cenjor Espanol C, Moreno-Parrado L, Ausina-Marquez V, Garcia-Esteban S, Artacho A, Lopez-Labrador FX, Mira A, Ferrer MD. Effect of oral antiseptics in reducing SARS-CoV-2 infectivity: evidence from a randomized double-blind clinical trial. Emerg Microbes Infect. 2022 Dec;11(1):1833-1842. doi: 10.1080/22221751.2022.2098059. PMID 35796097
- [Derived] Ferrer MD, Barrueco AS, Martinez-Beneyto Y, Mateos-Moreno MV, Ausina-Marquez V, Garcia-Vazquez E, Puche-Torres M, Giner MJF, Gonzalez AC, Coello JMS, Rueda IA, Auba JMV, Espanol CC, Velasco AL, Abad DS, Garcia-Esteban S, Artacho A, Lopez-Labrador X, Mira A. Clinical evaluation of antiseptic mouth rinses to reduce salivary load of SARS-CoV-2. Sci Rep. 2021 Dec 22;11(1):24392. doi: 10.1038/s41598-021-03461-y. PMID 34937855